CLINICAL TRIAL: NCT02251587
Title: The $Ensible Weight Program: An Intervention Tailored for Low Income Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeannine Goetz, PhD (Other)
Responsible Party: Sponsor-Investigator, Jeannine Goetz, PhD, Assistant Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001503
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Weight Management Program (Active Comparator): Participants will be given information on diet and exercise. Participants will attend meetings to discuss barriers to exercise and nutrition and ways to solve these problems. Participants will be given healthy snack ideas and planning tools.
  Interventions: Other: Standard Weight Management Program
- $ensible Weigh Program (Experimental): Participants will be given information on diet and exercise with an emphasis on food security. Participants will be provided with additional information on community resources such as those for food, transportation, and safe places to exercise. A weekly cooking demonstration will be provided using inexpensive ingredients and common food pantry items.
  Interventions: Other: Sensible Weigh Program

INTERVENTIONS:
Other: Standard Weight Management Program — Standard Diet program based on diet and exercise.
  Arms: Standard Weight Management Program
Other: Sensible Weigh Program — Weight loss program designed for low income women.
  Arms: $ensible Weigh Program

SUMMARY:
The purpose of this study is to learn if a weight loss program especially designed to address food insecurity is more effective compared to a standard weight loss program.

DETAILED DESCRIPTION:
Low income women are at greater risk of both obesity and food insecurity (not having consistent access to nutritious and adequate amounts of food). Most weight loss programs targeted at low income women do not focus on gaining skills and knowledge to reduce food insecurity.

Eligible participants will be randomized into one of two groups. The two groups will follow different weight management programs. One group will follow a standard weight management program. The other group with follow the investigations program, the $ensible Weigh Program. Participation in the study will last about 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented low income
* Body Mass Index (BMI) >25.0 kg/m2
* Must speak and understand English
* Able to attend intervention sessions and have access to telephone

Exclusion Criteria:

* Report serious medical risk such as insulin-dependent diabetes, cancer, recent cardiac event
* Currently or planning to become pregnant during the intervention
* Have no control over food purchases or choices
* Report participation in a weight reduction program involving diet or PA within past 6 months
* Report symptomology of an eating disorder
* Report adherence to specialized diet regimes, i.e., multiple food allergies, vegetarian, Atkins, macrobiotic, etc.

Ages: 21 Months to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementing weight management program | 9 Months
  Feasibility assessed by participant retention, participant attendance at study related visits, and participant satisfaction.

SECONDARY OUTCOMES:
Change in weight | Change from Baseline to Month 3
  Change in weight during the weight loss phase
Change in weight | Change from Month 3 to Month 9
  Change in weight during the weight management phase
Change in diet quality | Change from Baseline to Month 3
  Change during the weight loss phase. Change will be measured based on questions answered about participant's diet quality. Changes measured based on lower percentage of calories from fat and increased consumption of fruits, vegetables and whole grains.
Change in diet quality | Change from Month 3 to Month 9
  Change during the weight management phase. Change will be measured based on questions answered about participant's diet quality. Changes measured based on lower percentage of calories from fat and increased consumption of fruits, vegetables and whole grains.
Change in food security status | Change from Baseline to Month 3
  Change during the weight loss phase. Change will be measured based upon responses to the US Household Food Security Questionnaire
Change in food security status | Change from Month 3 to Month 9
  Change during the weight maintenance phase. Change will be measured based upon responses to the US Household Food Security Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jeannine Goetz, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States